CLINICAL TRIAL: NCT06658717
Title: A Randomized, Double-Blind, Two-Arm, Placebo-Controlled Clinical Study to Assess the Effect of the Natural Orange Extract in Individuals With Gastrointestinal Discomfort
Brief Title: A Study to Assess the Effect of the Natural Orange Extract in Individuals With Gastrointestinal Discomfort
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HT/240501/CARD/GID
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-09

CONDITIONS: Gut Health

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, two-arm, placebo-controlled clinical study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: Investigational product (IP) (Experimental): One capsule to be taken with breakfast orally once a day
  Interventions: Dietary Supplement: Investigational product (IP): Natural orange extract
- Placebo: Microcrystalline cellulose (MCC) (Placebo Comparator): One capsule to be taken with breakfast orally once a day
  Interventions: Dietary Supplement: Group II: Placebo: Microcrystalline cellulose (MCC)

INTERVENTIONS:
Dietary Supplement: Investigational product (IP): Natural orange extract — Strength: 500 mg Dose regimen: One capsule to be taken with breakfast orally once a day
  Arms: Group I: Investigational product (IP)
Dietary Supplement: Group II: Placebo: Microcrystalline cellulose (MCC) — Strength: 500 mg Dose regimen: One capsule to be taken with breakfast orally once a day
  Arms: Placebo: Microcrystalline cellulose (MCC)

SUMMARY:
A Randomized, Double-Blind, Two-Arm, Placebo-Controlled Clinical Study to assess the Effect of the Natural Orange Extract in Individuals with Gastrointestinal Discomfort

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Two-Arm, Placebo-Controlled Clinical Study to assess the Effect of the Natural Orange Extract in Individuals with Gastrointestinal Discomfort

ELIGIBILITY:
Inclusion Criteria:

1. Individuals willing to give written informed consent form voluntarily to participate in the study
2. Healthy males and females of age between 18-65 years.
3. Individuals with a Body Mass Index (BMI) between 18.5-29.9 kg/m2 (both values included).
4. Individuals with a history of GI discomfort, associated with changes in the frequency and form of stools for the last 3 months, with symptom onset at least 6 months.
5. Individuals with complaints of loose or watery stools, occurring in more than 25% of stools for the last 3 months.
6. Individuals with consistent and stable body weight in the last 3 months prior to screening (less than 5% self-reported change).
7. Individuals with a baseline score of less than or equal to 55 for the digestive domain score of the Gastrointestinal Quality of Life Index (GIQLI).
8. Individuals with Fasting Blood Glucose (FBG) less than equal to 125 mg/dl.
9. Individuals with systolic blood pressure (SBP) less than 140 and/or diastolic blood pressure (DBP) less than 90 mm Hg.
10. Individuals willing to avoid consumption of citrus-based products during the entire study duration.
11. Individuals willing to follow all the study procedures and follow-up visits as per protocol.

Exclusion Criteria:

1. Individuals diagnosed with diabetes mellitus and are on active medication.
2. Individuals diagnosed with hypertension and are on active medication.
3. Individuals with thyroid dysfunction as assessed by Thyroid Stimulating Hormone (TSH) less than or equal to 0.4 or more than or equal to 5.0 mIU/L will be excluded.
4. Individuals with a history and/or presence of acute or chronic significant GI disease or digestion/absorption disorders (e.g., Irritable bowel syndrome, inflammatory bowel disease, infectious diarrhea, coeliac disease, Clostridium difficile colitis, malabsorption, pancreatitis, disorders in digestive tract motility, gluten enteropathy, etc).
5. Individuals with a history of autoimmune disorders.
6. Individuals with major gastric, hepatic, biliary, pancreatic, or intestinal surgery within the last 6 months prior to screening or planned during the study (appendectomy, haemorrhoidectomy, or polypectomy allowed as long as occurred more than 3 months prior to screening; uncomplicated laparoscopic or open cholecystectomy is allowed if no history of post-operative biliary tract pain and surgery occurred more than 3 months prior to screening).
7. Any other relevant serious organ or systemic diseases (e.g., cardiovascular, respiratory, liver, renal, neurological disease, etc).
8. Individuals with a history of malignancy within last five years.
9. Use of immunosuppressive drugs within 3 months prior to the screening.
10. Use of oral corticosteroids within 1 month prior to the screening.
11. Excessive alcohol drinking (For men, consuming five or more drinks on any day or 15 or more per week; for women, consuming four or more on any day or 8 or more drinks per week). One unit of alcohol is equal to 45 ml of hard liquor, 150 ml of wine or a pint of beer.
12. Individuals with a history of/known allergies to citrus fruits or citrus-based products.
13. Individuals taking any antibiotics in the past 4 weeks and during the study.
14. Individuals who are on regular intake of laxatives in the past 1 month prior to the screening.
15. Individuals taking any dietary supplements, and medication for any gastrointestinal or metabolic disease (peptic ulcer, IBS, type-II diabetes, atherosclerosis, etc.)
16. Individuals taking any hormones for any gastrointestinal or metabolic disease within 3 months prior to screening.
17. Individuals taking any probiotics, prebiotics, post-biotics or synbiotics within 3 months prior to the screening.
18. History of smoking or currently smoking.
19. Individuals with gluten and/or lactose intolerance.
20. Females who are pregnant/lactating or planning to be pregnant.
21. Individuals who have participated in another clinical study(ies) with an IP within 90 days before screening, or who plan to participate in another study during the study period.
22. Any other conditions, which in the opinion of the investigator may jeopardize the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of the IP on gastrointestinal digestion symptoms as assessed by the change in digestive domain scores of the Gastrointestinal Quality of Life Index (GIQLI) compared to baseline and placebo. | Day 0, Day 45, Day 90.
  GIQLI is a validated tool suitable for assessing health-related quality of life (QOL) in clinical studies of individuals with gastrointestinal conditions and in routine clinical settings. It evaluates both generic and specific upper and lower gastrointestinal symptoms through 36 items. These questions are grouped into five domains: core symptoms (10 items), physical items (6 items), psychological items (6 items), social items (2 items) and disease-specific items (8 items).
  The GIQLI total cumulative score for the digestive domain ranges from 0 to 72, with higher scores indicating better gastrointestinal function and quality of life in the context of digestive symptoms

SECONDARY OUTCOMES:
To assess the effect of IP on the following compared to baseline and placebo Gastrointestinal quality of Life as assessed by GIQLI | Day 0, Day 45, Day 90
  GIQLI is a validated tool suitable for assessing health-related quality of life (QOL) in clinical studies of individuals with gastrointestinal conditions and in routine clinical settings. It evaluates both generic and specific upper and lower gastrointestinal symptoms through 36 items. These questions are grouped into five domains: core symptoms (10 items), physical items (6 items), psychological items (6 items), social items (2 items) and disease-specific items (8 items).
  The GIQLI total cumulative score for the digestive domain ranges from 0 to 72, with higher scores indicating better gastrointestinal function and quality of life in the context of digestive symptoms
To assess the effect of IP on the following compared to baseline and placebo Stool consistency as assessed by the Bristol Stool Form Scale (BSFS) | Day 0, Day 45, Day 90
  The Bristol Stool Form Scale (BSFS) is a 7-point ordinal scale of stool types extensively used in clinical and research settings that classify feces into seven groups
To assess the effect of IP on the following compared to baseline and placebo on Percentage responders as assessed by the change in the frequency of BSFS stool types 6 & 7 | Day 0, Day 45, Day 90
  The Bristol Stool Form Scale (BSFS) is a 7-point ordinal scale of stool types extensively used in clinical and research settings that classify feces into seven groups
To assess the effect of IP on the following compared to baseline and placebo on Gastrointestinal symptoms as assessed by the Gastrointestinal Symptoms Rating scale (GSRS) | Day 0, Day 45, Day 90
  The GSRS is a self-reported questionnaire for GI discomfort. The questions in this scale ask about the severity of a wide range of gastrointestinal symptoms of an individual during the past week. Questions are to be rated on a Likert scale ranging from no discomfort at all (0) to very severe discomfort (3). A total score is calculated by summing the ratings provided on all questions
To assess the effect of IP on the compared to baseline and placebo Intestinal permeability as assessed by serum levels of Lipopolysaccharide binding protein (LBP) | Day 0 & Day 90
  LPS is detected throughout the body by a specific protein called Lipopolysaccharide binding protein (LBP). LBP then initiates the immune response by presenting LPS to cell surface pattern recognition receptors membrane-bound CD14 (mCDC14) and toll-like receptor-4 (TLR4).
To assess the effect of IP on the compared to baseline and placebo on Inflammation as assessed by Interleukin-6 (IL-6), Interleukin-10 (IL-10) and Tumor Necrosis Factor-alpha (TNF-α) | Day 0 & Day 90
  Inflammation serves as a natural defensive reaction of the innate immune system triggered by various harmful agents such as microorganisms, trauma, necrosis, chemicals, immune responses, or metabolic stress.
  The acceptable ranges proposed are as follows: IL-6 (Not detectable to 50 pg/ml), IL-10 (Not detectable to 8 pg/ml), and TNF-α (2 to 20 pg/ml)
To assess the effect of IP on the compared to baseline and placebo on Intestinal inflammation as assessed by fecal calprotectin. | Day 0 & Day 90
  The fecal calprotectin a highly sensitive marker for detecting inflammation associated with GI disorders. The concentration of fecal calprotectin correlates well with the severity of intestinal inflammation,The fecal calprotectin range was found to be 18-37 μg /g in IBS individuals
To assess the effect of IP on the compared to baseline and placebo on Microbial metabolic activity as assessed by fecal short-chain fatty acids (SCFA) [Acetate, Butyrate and Propionate] | Day 0 & Day 90
  SCFAs exert beneficial effects on gut health through various mechanisms. They help maintain intestinal barrier integrity, promote mucus production, and possess anti-inflammatory properties, thereby contributing to overall GI well-being.
  These SCFAs range from 20 to 140 mM in the gut, with higher concentrations found in the proximal colon (70-140 mM) and lower concentrations in the distal colon (20-70 mM) and distal ileum (20-40 mM).
To assess the effect of IP on the compared to baseline and placebo on The gut microbiome as assessed by Next Generation Sequencing (NGS) | Day 0 & Day 90
  NGS allows for a more comprehensive analysis of complex microbial communities compared to traditional culture-based methods. The declining costs associated with NGS have further propelled its widespread adoption in microbiome research. NGS has proven particularly advantageous in elucidating the intricate relationship between the microbiome and various conditions.NGS will be assessed on day 0 and day 90

CONTACTS AND LOCATIONS:
Locations (3):
- India (3):
  - Pawna Hospital, Pune, Maharashtra
  - Shree Samarth Hospital, Pune, Maharashtra
  - Shivam Hospital, Thane, Maharashtra

IPD SHARING:
Plan to Share IPD: No